CLINICAL TRIAL: NCT02565914
Title: A Phase 3, Open-label, Rollover Study to Evaluate the Safety and Efficacy of Long Term Treatment With VX-661 in Combination With Ivacaftor in Subjects Aged 12 Years and Older With Cystic Fibrosis, Homozygous or Heterozygous for the F508del-CFTR Mutation
Brief Title: A Study to Evaluate the Safety and Efficacy of Long Term Treatment With VX-661 in Combination With Ivacaftor in Participants With Cystic Fibrosis Who Have an F508del-CFTR Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX14-661-110; 2014-004827-29 (EudraCT Number)
Record Dates: First submitted 2015-09-18; First posted 2015-10-01 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor, ivacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TEZ/IVA (Experimental): Part A: Participants who received either TEZ/IVA, IVA monotherapy or Placebo in parent studies 103,106,107,108,109 and 111 were administered TEZ 100 milligram (mg)/IVA 150 mg fixed-dose tablet in the morning and IVA 150 mg mono tablet in the evening for 96 weeks.
  Part B: Participants who received either TEZ/IVA, IVA monotherapy or Placebo in parent studies 106,108,109,112 and 114 were administered TEZ 100 mg/IVA 150 mg fixed-dose tablet in the morning and IVA 150 mg mono tablet in the evening for 96 weeks.
  Part C: Participants who received TEZ/IVA, IVA monotherapy or Placebo in parent studies 106,108, and 114 were administered TEZ 100 mg/IVA 150 mg fixed dose tablet in the morning and IVA 150 mg mono tablet in the evening for 192 weeks.
  Interventions: Drug: TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: TEZ/IVA — Fixed dose tablet for oral administration.
  Other Names: VX-661/VX-770; tezacaftor/ivacaftor
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
This is a Phase 3, multicenter, open-label, 3-part rollover study in subjects with CF who are homozygous or heterozygous for the F508del-CFTR mutation and who participated in studies VX13-661-103 (Study 103, NCT02070744), VX14-661-106 (Study 106, NCT02347657), VX14-661-107 (Study 107, NCT02516410), VX14-661-108 (Study 108, NCT02392234), VX14-661-109 (Study 109, NCT02412111), VX14-661-111 (Study 111, NCT02508207), VX15-661-112 (NCT02730208), and VX16-661-114 (NCT03150719). The study is designed to evaluate the safety and efficacy of long-term treatment of VX-661 in combination with ivacaftor.

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Participants entering the Treatment Cohort must meet all of the following criteria:
* Elect to enroll in the Treatment Cohort
* Completed study drug Treatment Period in a parent study (NCT02070744, NCT02347657, NCT02516410, NCT02392234, NCT02412111) or study drug treatment and the Safety Follow up Visit for participants from NCT02508207.
* Willing to remain on a stable CF regimen through the Safety Follow-up Visit.
* Participants re-enrolling in the Part A Treatment Cohort must meet all of the following criteria:

  * Previously received at least 4 weeks of study drug before discontinuing in Part A of Study NCT02565914 to participate in another qualified Vertex study.
  * Completed the last required visit of another qualified Vertex study before or during the Returning Visit in Part A Study NCT02565914.
* Participants entering the Part A Observational Cohort must meet the following criteria:

  * <18 years of age (age on the date of informed consent/assent in the parent study)
  * Completed study drug Treatment Period in a parent study or study drug treatment and the Safety Follow up Visit for subjects from NCT02508207, but do not elect to enroll in the NCT02565914 Treatment Cohort; or
  * Received at least 4 weeks of study drug treatment and completed visits up to the last scheduled visit of the Treatment Period of a parent study (and the Safety Follow up Visit for participants from NCT02508207), but do not meet eligibility criteria for enrollment into the Treatment Cohort

Part B:

Participants who meet all of the following inclusion criteria will be eligible for Part B.

* Did not withdraw consent from the parent study or Part A of Study NCT02565914.
* Completed study drug treatment during the Treatment Period in Part A of - Willing to remain on a stable CF medication (and supplement) regimen through the 96 week visit of Study NCT02565914.

Participants re enrolling in Part B must meet all of the following criteria:

* Previously received at least 4 weeks of study drug before discontinuing Study NCT02565914 to participate in another qualified Vertex study, which is defined as a Vertex study of investigational CFTR modulators that allows participation of participants in Study NCT02565914.
* Completed the last required visit of another qualified Vertex study before or during the Returning Visit in Part B.
* Willing to remain on a stable CF medication (and supplement) regimen through the 96 week visit in Part B.

Part C:

* Participants who meet all of the following inclusion criteria will be eligible for Part C.
* Did not withdraw consent from Part B of Study NCT02565914.
* Completed study drug treatment during Part B of NCT02565914.
* Willing to remain on a stable CF medication (and supplement) regimen through the 96 week visit of Part C.

Exclusion Criteria:

* History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk to the subject.
* Pregnant and nursing females.
* Sexually active subjects of reproductive potential who are not willing to follow the contraception requirements.
* History of drug intolerance in the parent study that would pose an additional risk to the subject.
* Participation in an investigational drug trial (including studies investigating VX-661/ivacaftor or lumacaftor/ivacaftor) other than the parent studies of NCT02565914 or other eligible Vertex studies investigating VX-661 in combination with ivacaftor, or use of a commercially available CFTR modulator.

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1131 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (154):
- United States (69):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Long Beach, California
  - Los Angeles, California
  - Oakland, California
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - Aurora, Colorado
  - Denver, Colorado
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Glenview, Illinois
  - Niles, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Long Branch, New Jersey
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Buffalo, New York
  - New Hyde Park, New York
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Sioux Falls, South Dakota
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Spokane, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Australia (4):
  - Chermside
  - Melbourne
  - South Brisbane
  - Westmead
- Austria (3):
  - Graz
  - Innsbruck
  - Salzburg
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Canada (5):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Halifax
  - Montreal
  - Québec
- Copenhagen, Denmark
- France (10):
  - Benite Cedex
  - Bordeaux
  - Bron
  - Lille
  - Marseille
  - Montpellier
  - Paris
  - Rennes
  - Roscoff
  - Rouen
- Germany (12):
  - Berlin
  - Bochum
  - Erlangen
  - Essen
  - Frankfurt
  - Giesen
  - Hannover
  - Heidelberg
  - Jena
  - München
  - Tübingen
  - Würzburg
- Ireland (3):
  - Cork
  - Dublin
  - Limerick
- Israel (5):
  - Haifa, NAP
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Litwinsky
- Italy (10):
  - Ancona
  - Genova
  - Milan
  - Orbassano
  - Palermo
  - Potenza
  - Roma
  - Rome
  - Torino
  - Verona
- Netherlands (5):
  - Amsterdam
  - Heidelberglaan
  - Nijmegen
  - Rotterdam
  - The Hague
- Spain (5):
  - Barcelona
  - Madrid
  - Sabadell
  - Seville
  - Valencia
- Sweden (3):
  - Gothenburg
  - Stockholm
  - Uppsala
- Switzerland (2):
  - Bern
  - Zurich
- United Kingdom (14):
  - Leeds, West Yorkshire
  - Belfast
  - Birmingham
  - Exeter
  - Glasgow
  - Leeds
  - Liverpool
  - London
  - Manchester
  - Newcastle upon Tyne
  - Penarth
  - Sheffield
  - Southampton
  - Stoke-on-Trent

REFERENCES:
- [Derived] Flume PA, Biner RF, Downey DG, Brown C, Jain M, Fischer R, De Boeck K, Sawicki GS, Chang P, Paz-Diaz H, Rubin JL, Yang Y, Hu X, Pasta DJ, Millar SJ, Campbell D, Wang X, Ahluwalia N, Owen CA, Wainwright CE; VX14-661-110 study group. Long-term safety and efficacy of tezacaftor-ivacaftor in individuals with cystic fibrosis aged 12 years or older who are homozygous or heterozygous for Phe508del CFTR (EXTEND): an open-label extension study. Lancet Respir Med. 2021 Jul;9(7):733-746. doi: 10.1016/S2213-2600(20)30510-5. Epub 2021 Feb 10. PMID 33581080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 3 parts: Parts A, B, and C.
Pre-assignment Details: A total 1131 participants enrolled in the study (1044 in Part A, 464 in Part B and 204 in Part C).
Groups:
- TEZ/IVA: Part A: Participants who received either TEZ/IVA, IVA monotherapy or Placebo in parent studies 103,106,107,108,109 and 111 were administered TEZ 100 mg/IVA 150 mg fixed-dose tablet in the morning and IVA 150 mg mono tablet in the evening for 96 weeks.
  Part B: Participants who received either TEZ/IVA, IVA monotherapy or Placebo in parent studies 106, 108, 109, 112 and 114 were administered TEZ 100 mg/IVA 150 mg fixed-dose tablet in the morning and IVA 150 mg mono tablet in the evening for 96 weeks.
  Part C: Participants who received TEZ/IVA, IVA monotherapy or Placebo in parent studies 106, 108, and 114 were administered TEZ 100 mg/IVA 150 mg fixed dose tablet in the morning and IVA 150 mg mono tablet in the evening for 192 weeks.
Period: Part A (Up to 96 Weeks)
Arm/Group | TEZ/IVA
Started | 1044
Safety Set (Received at least 1 dose of TEZ/IVA) | 1042
Completed | 951
Not Completed | 93
Not completed — Adverse Event | 17
Not completed — Withdrawal of consent (not due to AE) | 25
Not completed — Lost to Follow-up | 12
Not completed — Death (not treatment emergent) | 1
Not completed — Other noncompliance | 6
Not completed — Physician Decision | 6
Not completed — Parent study termination by sponsor | 1
Not completed — Commercial drug available | 5
Not completed — Other | 18
Not completed — Enrolled, but did not receive study drug | 2
Period: Part B (Up to 96 Weeks)
Arm/Group | TEZ/IVA
Started | 464 (Out of 464 participants in Part B, 377 participants rolled over from Part A and 87 participants rolled over directly from parent studies.)
Safety Set (Received at least 1 dose of TEZ/IVA) | 463
Completed | 228
Not Completed | 236
Not completed — Physician Decision | 1
Not completed — Other | 1
Not completed — Enrolled, but did not receive study drug | 1
Not completed — Adverse Event | 4
Not completed — Sponsor Decision | 2
Not completed — Rolled over into another study | 25
Not completed — Withdrawal of consent (not due to AE) | 6
Not completed — Commercial drug is available for participant | 196
Period: Part C (Up to 192 Weeks)
Arm/Group | TEZ/IVA
Started | 204 (Out of 464 participants in Part B, 204 participants rolled over to Part C.)
Safety Set | 204
Completed | 7
Not Completed | 197
Not completed — Physician Decision | 5
Not completed — Adverse Event | 1
Not completed — Other non-compliance | 2
Not completed — Rolled over into another study | 11
Not completed — Withdrawal of consent (not due to AE) | 4
Not completed — Commercial drug is available for participant | 174

BASELINE CHARACTERISTICS:
Population: Baseline data is based on the parent study baseline, which is defined as the most recent non-missing measurements collected before the first dose of the study drug in the treatment period of parent studies. Baseline data is presented for all participants who signed informed consent and enrolled, or dosed, in Part A, Part B, or Part C, respectively in this study.
Arm/Group | TEZ/IVA
Number analyzed (Participants) | 1131
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The Baseline data were planned to be presented separately for Part A , Part B and Part C. Here "Number Analyzed" signifies participants who were evaluable for the specified part of the study.
  years
    Part A: number analyzed (Participants) | 1044
    Part A | 29.13 (12.00)
    Part B: number analyzed (Participants) | 464
    Part B | 29.61 (11.89)
    Part C: number analyzed (Participants) | 204
    Part C | 29.60 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A, Part B and Part C. Here "Number Analyzed" signifies participants who were evaluable for the specified part of the study.
  Participants
    Part A: number analyzed (Participants) | 1044
    Part A: Female | 505
    Part A: Male | 539
    Part B: number analyzed (Participants) | 464
    Part B: Female | 221
    Part B: Male | 243
    Part C: number analyzed (Participants) | 204
    Part C: Female | 89
    Part C: Male | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A , Part B and Part C. Here "Number Analyzed" signifies participants who were evaluable for the specified part of the study.
  Participants
    Part A: number analyzed (Participants) | 1044
    Part A: Hispanic or Latino | 25
    Part A: Not Hispanic or Latino | 1002
    Part A: Not collected per local regulations | 17
    Part B: number analyzed (Participants) | 464
    Part B: Hispanic or Latino | 6
    Part B: Not Hispanic or Latino | 437
    Part B: Not collected per local regulations | 21
    Part C: number analyzed (Participants) | 204
    Part C: Hispanic or Latino | 5
    Part C: Not Hispanic or Latino | 184
    Part C: Not collected per local regulations | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented separately for Part A , Part B and Part C. Here "Number Analyzed" signifies participants who were evaluable for the specified part of the study.
  Participants
    Part A: number analyzed (Participants) | 1044
    Part A: White | 1017
    Part A: Black or African American | 7
    Part A: Asian | 2
    Part A: American Indian or Alaska Native | 1
    Part A: Native Hawaiian or Other Pacific Islander | 0
    Part A: Not collected per local regulations | 11
    Part A: Other | 6
    Part B: number analyzed (Participants) | 464
    Part B: White | 447
    Part B: Black or African American | 1
    Part B: Asian | 2
    Part B: American Indian or Alaska Native | 0
    Part B: Native Hawaiian or Other Pacific Islander | 0
    Part B: Not collected per local regulations | 13
    Part B: Other | 1
    Part C: number analyzed (Participants) | 204
    Part C: White | 193
    Part C: Black or African American | 0
    Part C: Asian | 1
    Part C: American Indian or Alaska Native | 0
    Part C: Native Hawaiian or Other Pacific Islander | 0
    Part C: Not collected per local regulations | 10
    Part C: Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 100
Population: Safety Set was defined as all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: TEZ/IVA: Participants who received either TEZ/IVA, IVA monotherapy or Placebo in parent studies 103,106,107,108,109 and 111 were administered TEZ 100 mg/IVA 150 mg fixed-dose tablet in the morning and IVA 150 mg mono tablet in the evening for 96 weeks.
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 1042
Participants
  Participants with TEAEs | 995
  Participants with SAEs | 351

2. Primary Outcome: Part B: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs
Time Frame: Day 1 up to Week 100
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: TEZ/IVA: Participants who received either TEZ/IVA, IVA monotherapy or Placebo in parent studies 106, 108, 109, 112 and 114 were administered TEZ 100 mg/IVA 150 mg fixed-dose tablet in the morning and IVA 150 mg mono tablet in the evening for 96 weeks.
Arm/Group | Part B: TEZ/IVA
Number analyzed (Participants) | 463
Participants
  Participants with TEAEs | 427
  Participants with SAEs | 136

3. Primary Outcome: Part C: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 196
Population: Safety set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part C: TEZ/IVA: Participants who received TEZ/IVA, IVA monotherapy or Placebo in parent studies 106, 108, and 114 were administered TEZ 100 mg/IVA 150 mg fixed dose tablet in the morning and IVA 150 mg mono tablet in the evening for 192 weeks.
Arm/Group | Part C: TEZ/IVA
Number analyzed (Participants) | 204
Participants
  Participants with TEAEs | 168
  Participants with SAEs | 44

4. Secondary Outcome: Part A: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) for 106/110 Efficacy Set
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 106 and TEZ/IVA in current study 110) and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 106 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline except for Placebo-TEZ/IVA category, for which baseline was study 110 baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: The 106/110 efficacy set included all enrolled participants who received at least 1 dose of study drug in Part A and rolled over from parent study 106 and had pre-defined CFTR genotypes.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 459
percentage points
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 231
  Placebo-TEZ/IVA: Change at Week 96 | 2.1 [0.8 to 3.3]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 228
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 2.0 [0.7 to 3.2]

5. Secondary Outcome: Part A: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) for 108/110 Efficacy Set
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 108 and TEZ/IVA in current study 110); IVA-TEZ/IVA category (participants who received IVA monotherapy in parent study 108 and TEZ/IVA in current study 110); and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 108 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: The 108/110 efficacy set included all enrolled participants who received at least 1 dose of study drug in Part A and rolled over from parent study 108 and had pre-defined CFTR genotypes.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 226
percentage points
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 80
  Placebo-TEZ/IVA: Change at Week 96 | 4.1 [2.2 to 6.0]
  IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 70
  IVA-TEZ/IVA: Change at Week 96 | 6.7 [4.7 to 8.7]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 76
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 7.5 [5.6 to 9.4]

6. Secondary Outcome: Part A: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) for 103/110 Efficacy Set
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Data are reported for TEZ/IVA-TEZ/IVA group (participants who received TEZ/IVA in both parent study 103 and in current study 110). Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: The 103/110 efficacy set included all enrolled participants who received at least 1 dose of study drug in Part A and rolled over from parent study 103 and had pre-defined CFTR genotypes.
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 23
percentage points | 2.7 (10.0)

7. Secondary Outcome: Part A: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) for 111/110 Efficacy Set
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 111 and TEZ/IVA in current study 110) and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 111 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: The 111/110 efficacy set included all enrolled participants who received at least 1 dose of study drug in Part A and rolled over from parent study 111 and had pre-defined CFTR genotypes.
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 33
percentage points
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 7
  Placebo-TEZ/IVA: Change at Week 96 | 4.1 (10.2)
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 26
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 2.6 (6.6)

8. Secondary Outcome: Part A: Relative Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) for 106/110 Efficacy Set
Description: as for outcome 4
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 459
percent change
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 231
  Placebo-TEZ/IVA: Change at Week 96 | 4.3 [2.1 to 6.5]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 228
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 4.2 [2.0 to 6.4]

9. Secondary Outcome: Part A: Relative Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) for 108/110 Efficacy Set
Description: as for outcome 5
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 226
percent change
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 80
  Placebo-TEZ/IVA: Change at Week 96 | 7.9 [4.7 to 11.1]
  IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 70
  IVA-TEZ/IVA: Change at Week 96 | 11.6 [8.2 to 15.0]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 76
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 13.0 [9.7 to 16.2]

10. Secondary Outcome: Part A: Relative Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) for 103/110 Efficacy Set
Description: as for outcome 6
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 23
percent change | 6.4 (21.1)

11. Secondary Outcome: Part A: Relative Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) for 111/110 Efficacy Set
Description: as for outcome 7
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 33
percent change
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 7
  Placebo-TEZ/IVA: Change at Week 96 | 6.1 (14.4)
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 26
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 5.2 (11.5)

12. Secondary Outcome: Part A: Number of Pulmonary Exacerbation (PEx) Events for 106/110 PEx Analysis Set
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms. Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 106 and TEZ/IVA in current study 110) and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 106 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline except for Placebo-TEZ/IVA category, for which baseline was study 110 baseline.
Time Frame: From Baseline up to Study 110 Week 96
Population: The 106/110 PEx analysis set included study 106 participants who received TEZ/IVA in Study 106 or Study 110.
Measure: Number; unit: PEx events
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 479
PEx events
  Placebo-TEZ/IVA: number analyzed (Participants) | 231
  Placebo-TEZ/IVA | 306
  TEZ/IVA-TEZ/IVA: number analyzed (Participants) | 248
  TEZ/IVA-TEZ/IVA | 423

13. Secondary Outcome: Part A: Number of Pulmonary Exacerbation (PEx) Events for 108/110 PEx Analysis Set
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms. Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 108 and TEZ/IVA in current study 110); IVA-TEZ/IVA category (participants who received IVA monotherapy in parent study 108 and TEZ/IVA in current study 110); and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 108 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline up to Week 96
Population: The 108/110 PEx analysis set included study 108 participants who received TEZ/IVA in Study 108 or Study 110.
Measure: Number; unit: PEx events
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 233
PEx events
  Placebo-TEZ/IVA: number analyzed (Participants) | 81
  Placebo-TEZ/IVA | 89
  IVA-TEZ/IVA: number analyzed (Participants) | 74
  IVA-TEZ/IVA | 51
  TEZ/IVA-TEZ/IVA: number analyzed (Participants) | 78
  TEZ/IVA-TEZ/IVA | 46

14. Secondary Outcome: Part A: Absolute Change in Body Mass Index (BMI) for 106/110 Efficacy Set
Description: BMI was defined as weight in kilogram (kg) divided by height in square meter (m^2). Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 106 and TEZ/IVA in current study 110) and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 106 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline except for Placebo-TEZ/IVA category, for which baseline was study 110 baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 459
kg/m^2
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 231
  Placebo-TEZ/IVA: Change at Week 96 | 0.47 [0.30 to 0.65]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 228
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 0.38 [0.20 to 0.55]

15. Secondary Outcome: Part A: Absolute Change in Body Mass Index (BMI) for 108/110 Efficacy Set
Description: BMI was defined as weight in kg divided by height in square meter (m^2). Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 108 and TEZ/IVA in current study 110); IVA-TEZ/IVA category (participants who received IVA monotherapy in parent study 108 and TEZ/IVA in current study 110); and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 108 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 226
kg/m^2
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 80
  Placebo-TEZ/IVA: Change at Week 96 | 1.07 [0.59 to 1.55]
  IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 70
  IVA-TEZ/IVA: Change at Week 96 | 0.96 [0.45 to 1.47]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 76
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 1.05 [0.56 to 1.55]

16. Secondary Outcome: Part A: Absolute Change in Body Mass Index (BMI) for 103/110 Efficacy Set
Description: BMI was defined as weight in kg divided by height in square meter (m^2). Data are reported for TEZ/IVA-TEZ/IVA group (participants who received TEZ/IVA in both parent study 103 and in current study 110). Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 23
kg/m^2 | 1.38 (1.73)

17. Secondary Outcome: Part A: Absolute Change in Body Mass Index (BMI) for Study 111/110 Efficacy Set
Description: BMI was defined as weight in kg divided by height in square meter (m^2). Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 111 and TEZ/IVA in current study 110) and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 111 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 33
kg/m^2
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 7
  Placebo-TEZ/IVA: Change at Week 96 | 1.59 (2.08)
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 26
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 0.26 (0.88)

18. Secondary Outcome: Part A: Absolute Change in BMI Z-score for 106/110 Efficacy Set
Description: The z-score is a statistical measure to describe whether a mean was above or below the standard. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 106 and TEZ/IVA in current study 110) and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 106 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline except for Placebo-TEZ/IVA category, for which baseline was study 110 baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: The 106/110 efficacy set included all enrolled participants <20 years of age at Screening who received at least 1 dose of study drug in Part A and rolled over from parent study 106 and had pre-defined CFTR genotypes.
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 93
z-score
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 44
  Placebo-TEZ/IVA: Change at Week 96 | 0.10 [-0.04 to 0.25]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 49
  TEZ/IVA-TEZ/IVA: Change at Week 96 | -0.14 [-0.28 to 0.00]

19. Secondary Outcome: Part A: Absolute Change in BMI Z-score for 108/110 Efficacy Set
Description: The z-score is a statistical measure to describe whether a mean was above or below the standard. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 108 and TEZ/IVA in current study 110); IVA-TEZ/IVA category (participants who received IVA monotherapy in parent study 108 and TEZ/IVA in current study 110); and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 108 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: The 108/110 efficacy set included all enrolled participants <20 years of age at Screening who received at least 1 dose of study drug in Part A and rolled over from parent study 108 and had pre-defined CFTR genotypes.
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 30
z-score
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 13
  Placebo-TEZ/IVA: Change at Week 96 | 0.11 [-0.32 to 0.54]
  IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 7
  IVA-TEZ/IVA: Change at Week 96 | 0.07 [-0.52 to 0.65]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 10
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 0.30 [-0.21 to 0.80]

20. Secondary Outcome: Part A: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score for 106/110 Efficacy Set
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 106 and TEZ/IVA in current study 110) and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 106 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline except for Placebo-TEZ/IVA category, for which baseline was study 110 baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 459
units on a scale
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 231
  Placebo-TEZ/IVA: Change at Week 96 | 1.7 [-0.6 to 4.0]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 228
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 3.0 [0.7 to 5.3]

21. Secondary Outcome: Part A: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score for 108/110 Efficacy Set
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 108 and TEZ/IVA in current study 110); IVA-TEZ/IVA category (participants who received IVA monotherapy in parent study 108 and TEZ/IVA in current study 110); and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 108 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 226
units on a scale
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 80
  Placebo-TEZ/IVA: Change at Week 96 | 10.3 [7.0 to 13.6]
  IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 70
  IVA-TEZ/IVA: Change at Week 96 | 11.2 [7.7 to 14.7]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 76
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 13.8 [10.3 to 17.2]

22. Secondary Outcome: Part A: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score for 103/110 Efficacy Set
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Data are reported for TEZ/IVA-TEZ/IVA group (participants who received TEZ/IVA in both parent study 103 and in current study 110). Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 23
units on a scale | 8.6 (12.1)

23. Secondary Outcome: Part A: Absolute Change in Body Weight for Study 106/110 Efficacy Set
Description: Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 106 and TEZ/IVA in current study 110) and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 106 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline except for Placebo-TEZ/IVA category, for which baseline was study 110 baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 459
kg
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 231
  Placebo-TEZ/IVA: Change at Week 96 | 2.0 [1.4 to 2.5]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 228
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 2.1 [1.5 to 2.6]

24. Secondary Outcome: Part A: Absolute Change in Body Weight for 108/110 Efficacy Set
Description: Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 108 and TEZ/IVA in current study 110); IVA-TEZ/IVA category (participants who received IVA monotherapy in parent study 108 and TEZ/IVA in current study 110); and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 108 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 226
kg
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 80
  Placebo-TEZ/IVA: Change at Week 96 | 3.5 [1.9 to 5.1]
  IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 70
  IVA-TEZ/IVA: Change at Week 96 | 3.5 [1.8 to 5.2]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 76
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 3.6 [2.0 to 5.2]

25. Secondary Outcome: Part A: Absolute Change in Body Weight for 103/110 Efficacy Set
Description: Data are reported for TEZ/IVA-TEZ/IVA group (participants who received TEZ/IVA in both parent study 103 and in current study 110). Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 23
kg | 4.0 (5.0)

26. Secondary Outcome: Part A: Absolute Change in Body Weight for 111/110 Efficacy Set
Description: Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 111 and TEZ/IVA in current study 110) and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 111 and in current study 110) as per pre-specified analysis plan. Baseline was defined as the parent study baseline.
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 33
kg
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 7
  Placebo-TEZ/IVA: Change at Week 96 | 4.2 (5.7)
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 26
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 0.6 (2.6)

27. Secondary Outcome: Part A: Absolute Change in Body Weight Z-score for 106/110 Efficacy Set
Description: as for outcome 18
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 18
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 93
z-score
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 44
  Placebo-TEZ/IVA: Change at Week 96 | 0.07 [-0.06 to 0.20]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 49
  TEZ/IVA-TEZ/IVA: Change at Week 96 | -0.06 [-0.19 to 0.07]

28. Secondary Outcome: Part A: Absolute Change in Body Weight Z-score for 108/110 Efficacy Set
Description: as for outcome 19
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 19
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 30
z-score
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 13
  Placebo-TEZ/IVA: Change at Week 96 | 0.15 [-0.25 to 0.55]
  IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 7
  IVA-TEZ/IVA: Change at Week 96 | 0.09 [-0.45 to 0.62]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 10
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 0.43 [-0.04 to 0.90]

29. Secondary Outcome: Part A: Absolute Change in Height Z-score for 106/110 Efficacy Set
Description: as for outcome 18
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 18
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 91
z-score
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 42
  Placebo-TEZ/IVA: Change at Week 96 | 0.01 [-0.08 to 0.11]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 49
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 0.13 [0.04 to 0.22]

30. Secondary Outcome: Part A: Absolute Change in Height Z-score for 108/110 Efficacy Set
Description: as for outcome 19
Time Frame: From Baseline at Study 110 Week 96
Population: as for outcome 19
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 30
z-score
  Placebo-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 13
  Placebo-TEZ/IVA: Change at Week 96 | -0.04 [-0.23 to 0.15]
  IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 7
  IVA-TEZ/IVA: Change at Week 96 | 0.20 [-0.05 to 0.45]
  TEZ/IVA-TEZ/IVA: Change at Week 96: number analyzed (Participants) | 10
  TEZ/IVA-TEZ/IVA: Change at Week 96 | 0.23 [0.00 to 0.46]

31. Secondary Outcome: Part A: Time-to-first Pulmonary Exacerbation (PEx) for 106/110 PEx Analysis Set
Description: Time-to-first pulmonary exacerbation was analyzed using Kaplan-Meier estimates and expressed in terms of event-free probability. PEx was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms. Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 106 and TEZ/IVA in current study 110) and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 106 and in current study 110) as per pre-specified analysis plan.
Time Frame: 96 weeks
Population: The 106/110 PEx analysis set included study 106 participants who received TEZ/IVA in Study 106 or Study 110.
Measure: Number (95% Confidence Interval); unit: event-free probability
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 479
event-free probability
  Placebo-TEZ/IVA: number analyzed (Participants) | 231
  Placebo-TEZ/IVA | 0.470 [0.402 to 0.535]
  TEZ/IVA-TEZ/IVA: number analyzed (Participants) | 248
  TEZ/IVA-TEZ/IVA | 0.438 [0.374 to 0.501]

32. Secondary Outcome: Part A: Time-to-first Pulmonary Exacerbation (PEx) for 108/110 PEx Analysis Set
Description: Time-to-first pulmonary exacerbation was analyzed using Kaplan-Meier estimates and expressed in terms of event-free probability. PEx was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms. Data are reported separately for Placebo-TEZ/IVA category (participants who received placebo in parent study 108 and TEZ/IVA in current study 110); IVA-TEZ/IVA category (participants who received IVA monotherapy in parent study 108 and TEZ/IVA in current study 110); and TEZ/IVA-TEZ/IVA category (participants who received TEZ/IVA in both parent study 108 and in current study 110) as per pre-specified analysis plan.
Time Frame: 96 weeks
Population: The 108/110 PEx analysis set included study 108 participants who received TEZ/IVA in Study 108 or Study 110.
Measure: Number (95% Confidence Interval); unit: event-free probability
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 233
event-free probability
  Placebo-TEZ/IVA: number analyzed (Participants) | 81
  Placebo-TEZ/IVA | 0.497 [0.383 to 0.601]
  IVA-TEZ/IVA: number analyzed (Participants) | 74
  IVA-TEZ/IVA | 0.493 [0.372 to 0.603]
  TEZ/IVA-TEZ/IVA: number analyzed (Participants) | 78
  TEZ/IVA-TEZ/IVA | 0.639 [0.519 to 0.737]

33. Secondary Outcome: Part A: Plasma Concentrations of TEZ, TEZ Metabolite (M1-TEZ), Ivacaftor (IVA) and Ivacaftor Metabolite (M1-IVA)
Time Frame: Week 24
Population: The Pharmacokinetic set included data for all participants who received TEZ/IVA treatment and met PK data inclusion and exclusion criteria.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Part A: TEZ/IVA
Number analyzed (Participants) | 853
nanogram/milliliter (ng/mL)
  VX-661 | 2070 (1390)
  M1-661 | 4580 (2080)
  IVA | 892 (700)
  M1-IVA | 1740 (1070)

34. Secondary Outcome: Part B: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline at Study 110 Week 96
Population: The efficacy set included all enrolled participants who received at least 1 dose of study drug in Part B and rolled over from parent studies and had pre-defined CFTR genotypes. It was performed on each of the CFTR mutation groups separately (F508del/F508del and F508del/Residual Function). Here, "Number Analyzed" signifies participants who were evaluable for the specific category of CFTR genotypes.
Measure: Mean (Standard Deviation); unit: percentage points
Arm/Group | Part B: TEZ/IVA
Number analyzed (Participants) | 181
percentage points
  F/F Mutation: number analyzed (Participants) | 132
  F/F Mutation | 1.7 (10.2)
  F/RF Mutation: number analyzed (Participants) | 49
  F/RF Mutation | 8.3 (8.6)

35. Secondary Outcome: Part B: Absolute Change in Body Mass Index (BMI)
Description: BMI was defined as weight in kilogram (kg) divided by height in square meter (m^2).
Time Frame: From Baseline at Week 96
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Part B: TEZ/IVA
Number analyzed (Participants) | 198
kg/m^2
  F/F Mutation: number analyzed (Participants) | 138
  F/F Mutation | 0.70 (1.45)
  F/RF Mutation: number analyzed (Participants) | 60
  F/RF Mutation | 1.84 (2.21)

36. Secondary Outcome: Part B: Absolute Change in BMI Z-score
Description: The z-score is a statistical measure to describe whether a mean was above or below the standard. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean.
Time Frame: From Baseline at Week 96
Population: The efficacy set included all enrolled participants who received at least 1 dose of study drug in Part B and rolled over from parent studies and had pre-defined CFTR genotypes. It was performed on each of the CFTR mutation groups separately (F508del/F508del and F508del/Residual Function).Here, "Number Analyzed" signifies participants who were evaluable for the specific category of CFTR genotypes.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Part B: TEZ/IVA
Number analyzed (Participants) | 27
z-score
  F/F Mutation: number analyzed (Participants) | 21
  F/F Mutation | -0.03 (0.71)
  F/RF Mutation: number analyzed (Participants) | 6
  F/RF Mutation | 0.21 (0.46)

37. Secondary Outcome: Part B: Number of Pulmonary Exacerbation (PEx) Events
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms.
Time Frame: From Baseline up to Week 96
Population: as for outcome 34
Measure: Number; unit: PEx events
Arm/Group | Part B: TEZ/IVA
Number analyzed (Participants) | 453
PEx events
  F/F Mutation: number analyzed (Participants) | 347
  F/F Mutation | 386
  F/RF Mutation: number analyzed (Participants) | 106
  F/RF Mutation | 94

ADVERSE EVENTS:
Time Frame: Day 1 Through Safety Follow-up Visit (up to Week 100 for Part A, up to Week 100 for Part B and up to Week 196 for Part C)
Arm/Group | Part A: TEZ/IVA | Part B: TEZ/IVA | Part C: TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 1/1042 | 0/463 | 0/204
Serious Adverse Events (participants affected / at risk) | 351/1042 | 136/463 | 44/204
Other Adverse Events (participants affected / at risk) | 938/1042 | 391/463 | 149/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: TEZ/IVA (N=1042) | Part B: TEZ/IVA (N=463) | Part C: TEZ/IVA (N=204)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Pituitary enlargement (Endocrine disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 0 | 0
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 8 | 3 | 0
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 12 | 3 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 4 | 3 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 2 | 0
Device related thrombosis (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Medical device site erythema (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Gallbladder rupture (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 2 | 3
Food allergy (Immune system disorders) | 1 | 0 | 0
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 2 | 0 | 0
Appendicitis (Infections and infestations) | 5 | 1 | 1
Atypical mycobacterial lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Atypical mycobacterial pneumonia (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 4 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 243 | 103 | 28
Influenza (Infections and infestations) | 7 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Lung infection (Infections and infestations) | 2 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 7 | 4 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 3 | 0 | 0
Salpingitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 1
Tonsillitis (Infections and infestations) | 2 | 0 | 0
Typhoid fever (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0
Vascular device infection (Infections and infestations) | 2 | 0 | 1
Anaesthetic complication cardiac (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ear injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Peroneal nerve injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 0 | 1
Bacterial test positive (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 7 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 1
Computerised tomogram thorax abnormal (Investigations) | 0 | 0 | 1
Forced expiratory volume decreased (Investigations) | 3 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Influenza A virus test positive (Investigations) | 1 | 0 | 0
Influenza B virus test positive (Investigations) | 1 | 1 | 0
Pulmonary function test decreased (Investigations) | 1 | 0 | 0
Respiratory syncytial virus test positive (Investigations) | 1 | 0 | 0
Urine amphetamine positive (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign male reproductive tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 2 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Quadrantanopia (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 5 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 1
Disruptive mood dysregulation disorder (Psychiatric disorders) | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 0
Suicide attempt (Psychiatric disorders) | 3 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 4 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Renal infarct (Renal and urinary disorders) | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 2 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 25 | 10 | 6
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Urticarial vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: TEZ/IVA (N=1042) | Part B: TEZ/IVA (N=463) | Part C: TEZ/IVA (N=204)
Abdominal pain (Gastrointestinal disorders) | 101 | 35 | 7
Abdominal pain upper (Gastrointestinal disorders) | 44 | 26 | 2
Constipation (Gastrointestinal disorders) | 69 | 24 | 8
Diarrhoea (Gastrointestinal disorders) | 105 | 27 | 5
Nausea (Gastrointestinal disorders) | 105 | 21 | 9
Vomiting (Gastrointestinal disorders) | 80 | 12 | 7
Fatigue (General disorders) | 100 | 23 | 7
Pyrexia (General disorders) | 135 | 40 | 20
Immunisation reaction (Immune system disorders) | 0 | 0 | 15
COVID-19 (Infections and infestations) | 0 | 1 | 18
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 444 | 202 | 87
Influenza (Infections and infestations) | 62 | 26 | 2
Nasopharyngitis (Infections and infestations) | 227 | 88 | 13
Rhinitis (Infections and infestations) | 55 | 28 | 5
Sinusitis (Infections and infestations) | 80 | 20 | 7
Upper respiratory tract infection (Infections and infestations) | 135 | 43 | 12
Viral upper respiratory tract infection (Infections and infestations) | 69 | 15 | 1
Aspartate aminotransferase increased (Investigations) | 53 | 7 | 0
Bacterial test positive (Investigations) | 48 | 28 | 11
Blood creatine phosphokinase increased (Investigations) | 76 | 3 | 0
Pulmonary function test decreased (Investigations) | 55 | 8 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 62 | 29 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 57 | 23 | 11
Headache (Nervous system disorders) | 146 | 47 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 374 | 112 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 99 | 28 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 167 | 64 | 25
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 77 | 7 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 136 | 39 | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 56 | 15 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 55 | 16 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 53 | 2 | 2
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 223 | 46 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT02565914/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT02565914/SAP_001.pdf